CLINICAL TRIAL: NCT03695770
Title: Evaluation of a New Malaria Control Strategy Amongst Gold Miners Working Illegally in French Guiana (Malakit)
Acronym: MALAKIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier de Cayenne (Other)
Collaborators: Dr Stephen Vreden (Foundation for Scientific Research Suriname : SWOS) (Unknown); Oswaldo Cruz Foundation (Other); Dr Maylis Douine (Centre Hospitalier de Cayenne) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MALAKIT
Record Dates: First submitted 2018-09-28; First posted 2018-10-04 (Actual); Last update posted 2021-05-20 (Actual); Status verified 2021-05

CONDITIONS: Malaria; Public Health
MeSH Terms: conditions — Malaria | interventions — Receptor Protein-Tyrosine Kinases

STUDY DESIGN:
Intervention Model Description: before/after study design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- target population (Experimental): All the target population should be included in the experimental arm
  Interventions: Other: kit for self-diagnosis and self-treatment

INTERVENTIONS:
Other: kit for self-diagnosis and self-treatment — distribution of kits for malaria self-diagnosis and self-treatment after a training by health facilitators

SUMMARY:
Illegal gold miners in French Guiana, a French overseas territory ('département') located in Amazonia, often carry malaria parasites (up to 46.8%). While the Guiana Shield Region aims at malaria elimination, the high prevalence of Plasmodiumin this hard-to-reach population in conjunction with frequent incorrect use of artemisinin-based anti-malarials could favor the emergence of resistant parasites. Due to geographical and regulatory issues in French Guiana, usual malaria control strategies cannot be implemented in this particular context.Therefore, new strategies targeting this specific population in the forest are required.

Numerous discussions among health institutions and scientific partners from French Guiana, Brazil and Suriname have led to an innovative project based on the distribution of kits for self-diagnosis and self-treatment of Plasmodium infections. The kit-distribution will be implemented at "resting sites", which are areas across the border of French Guiana regularly frequented by gold miners. The main objective is to increase the appropriate use and complete malaria treatment after a positive malaria diagnosis with a rapid test, which will be evaluated with before-and-after cross-sectional studies. Monitoring indicators will be collected from health mediators at the time of kit distribution and during subsequent visits, and from illegal gold miners themselves, through a smartphone application. The project funding is multisource, including Ministries of Health of the three countries, WHO/PAHO, and the European Union.

DETAILED DESCRIPTION:
Background Despite a decrease in the number of cases reported to CIRE "Cellule de l'Institut de Veille Sanitaire", an interregional epidemiological surveillance center, malaria affects many gold miners working illegally in French Guiana. The ORPAL study carried out by CIC "Centre d'Investigation Clinique" (clinical investigation center) in 2015, showed that the prevalence of Plasmodium in illegal gold miners was 22.3%, of which 84% were asymptomatic. Self-medication practices are very common (52.4%) using artemisinin derivatives.

Key issues identified:

* The mobile population of workers in illegal gold mining sites is particularly affected by malaria due to their living and working conditions and as such represents a reservoir of transmission.
* Their undocumented irregular status and difficult access to health centers makes care from health professionals rare or belated.
* The use of inadequate drugs, without prior diagnosis and with improper compliance, mainly due to the high cost of treatment on the black market, is common. These non-recommended practices contribute to the risk of emergence of ACT resistance.
* Knowledge of the disease by illegal gold miners (causes, symptoms, preventive measures and treatment) remains insufficient.

Considering the problems, the identified need is to ensure sufficient intervention coverage of appropriate and rapid care, amongst the malaria "reservoir" population, in order to reduce:

* Malaria transmission and ACT non-compliance;
* The ensuing risk of P. falciparum resistance to ACT;
* The morbidity and mortality of illegal workers in gold-mining sites;

The working hypothesis is:

The free distribution of self-diagnosis and self-treatment kits, together with appropriate training / information, at "resting sites", Brazil and Suriname, would be a strategy relevant to the specific context of French Guiana, and would respond to the identified need.

Objectives This study aims to assess a new malaria control strategy targeting gold miners working illegally in French Guiana, based on the distribution of self-diagnosis kits and self-treatment against P. falciparum in cross-border areas.

* Main objective Increase the part of illegal gold miners in French Guiana who take ACT entirely after a positive rapid diagnostic test.
* Secondary objectives

  * Improve the use of anti-malarial treatments against P. falciparum appropriately and in compliance with WHO recommendations.
  * Reduce the prevalence of malaria among illegal gold miners in French Guiana.
  * Increase the part of illegal gold miners in French Guiana who:

    * Know malaria, its causes, the symptoms and protection measures.
    * Have a positive attitude towards recommended prevention measures, the use of adequate anti-malarial treatment, and adherence to treatment.
    * Report applying good preventive practices.

Project implementation:

This project will be carried out in cooperation with Brazil, Suriname and France. It is divided into 2 sections:

* Part 1: Implementation and monitoring of the intervention Distribution of self-diagnosis and self-treatment kits to people working illegally at gold-mining sites in French Guiana, along with the provision of training. This distribution will take place at resting sites by trained facilitators. Proactive digital collection of data will be conducted by these facilitators and via gold miners themselves through a mobile application.
* Part 2: Evaluation of the intervention The final evaluation of the project will be carried out in a cross-sectional study "Orpal bis", with a questionnaire on knowledge, attitudes and practices and blood sampling to measure the prevalence of Plasmodium carriers before / after the intervention. The same study (Orpal) was carried out in 2015 along the Surinamese border, and will be carried out before implementation along the Brazilian border.

Therefore, it will be a pre-post evaluation. Depending on the results, the sustainability of the action will be determined by the Health Authorities.

Duration As a pilot project, the inclusion period for which the data will be processed in the view of determining the potential sustainability is 12 months. The length of the results capitalizing is estimated to be 6 months, during which the intervention will be maintained, in order to avoid any useless gap. Therefore, the total duration of the pilot phase is 18 months.

ELIGIBILITY:
Inclusion Criteria:

* over 15 years-old
* working or accompanying someone working in illegal gold mining in French Guiana
* agreing to take part of the study
* to have parents authorization if age between 15 and 17 ;
* capable of performing a self-RDT during the training (validation by the facilitator);

Exclusion Criteria:

* refusing to participate in the study ;
* under 15 years old ;
* no parents authorization ;
* weighing less than 35 kg ;
* who has not been able to perform a self-RDT during the training (invalidation by the facilitator).

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 3733 (Actual)
Dates: Start 2018-04-16 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
KAP Questionnaire | 12 months
  change the part of illegal gold miners in French Guiana who take a correct antimalarial treatment (with artemisinin-combined therapy) with a good adherence and after a positive rapid diagnostic test.

SECONDARY OUTCOMES:
malaria prevalence | 12 months
  change PCR-Plasmodium prevalence amongst gold miners working illegally in French Guiana
KAP questionnaire | 12 months
  change the use of protection measures against mosquitoes

CONTACTS AND LOCATIONS:
Locations (2):
- Fondation Oswaldo Cruz, Rio de Janeiro, Brazil
- Foundation for Scientific Research Suriname (SWOS), Paramaribo, Suriname

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Douine M, Sanna A, Galindo M, Musset L, Pommier de Santi V, Marchesini P, Magalhaes ED, Suarez-Mutis M, Hiwat H, Nacher M, Vreden S, Garancher L. Malakit: an innovative pilot project to self-diagnose and self-treat malaria among illegal gold miners in the Guiana Shield. Malar J. 2018 Apr 10;17(1):158. doi: 10.1186/s12936-018-2306-5. PMID 29631588
- [Background] Douine M, Lazrek Y, Blanchet D, Pelleau S, Chanlin R, Corlin F, Hureau L, Volney B, Hiwat H, Vreden S, Djossou F, Demar M, Nacher M, Musset L. Predictors of antimalarial self-medication in illegal gold miners in French Guiana: a pathway towards artemisinin resistance. J Antimicrob Chemother. 2018 Jan 1;73(1):231-239. doi: 10.1093/jac/dkx343. PMID 29045645
- [Background] Douine M, Musset L, Corlin F, Pelleau S, Pasquier J, Mutricy L, Adenis A, Djossou F, Brousse P, Perotti F, Hiwat H, Vreden S, Demar M, Nacher M. Prevalence of Plasmodium spp. in illegal gold miners in French Guiana in 2015: a hidden but critical malaria reservoir. Malar J. 2016 Jun 9;15:315. doi: 10.1186/s12936-016-1367-6. PMID 27277831
- [Background] Pommier de Santi V, Djossou F, Barthes N, Bogreau H, Hyvert G, Nguyen C, Pelleau S, Legrand E, Musset L, Nacher M, Briolant S. Malaria Hyperendemicity and Risk for Artemisinin Resistance among Illegal Gold Miners, French Guiana. Emerg Infect Dis. 2016 May;22(5):903-6. doi: 10.3201/eid2205.151957. PMID 27089004
- [Background] van Eer ED, Bretas G, Hiwat H. Decreased endemic malaria in Suriname: moving towards elimination. Malar J. 2018 Jan 30;17(1):56. doi: 10.1186/s12936-018-2204-x. PMID 29378594
- [Background] Musset L, Pelleau S, Girod R, Ardillon V, Carvalho L, Dusfour I, Gomes MS, Djossou F, Legrand E. Malaria on the Guiana Shield: a review of the situation in French Guiana. Mem Inst Oswaldo Cruz. 2014 Aug;109(5):525-33. doi: 10.1590/0074-0276140031. Epub 2014 Aug 13. PMID 25184998
- [Derived] Longchamps C, Galindo MS, Lambert Y, Sanna A, Mutricy L, Garancher L, Adenis A, Nacher M, Suarez-Mutis M, Cairo H, Hiwat H, Vreden S, Douine M. Impact of Malakit intervention on perceptions, knowledge, attitudes, and practices related to malaria among workers in clandestine gold mines in French Guiana: results of multicentric cross-sectional surveys over time. Malar J. 2022 Dec 28;21(1):397. doi: 10.1186/s12936-022-04391-4. PMID 36577968
- [Derived] Lambert Y, Galindo M, Suarez-Mutis M, Mutricy L, Sanna A, Garancher L, Cairo H, Hiwat H, Bordalo Miller J, Gomes JH, Marchesini P, Adenis A, Nacher M, Vreden S, Douine M. Tailoring Mobile Data Collection for Intervention Research in a Challenging Context: Development and Implementation in the Malakit Study. JMIR Form Res. 2022 Jun 16;6(6):e29856. doi: 10.2196/29856. PMID 35708763
- [Derived] Galindo MS, Lambert Y, Mutricy L, Garancher L, Miller JB, Gomes JH, Sanna A, Peterka C, Cairo H, Hiwat H, Adenis A, Nacher M, Suarez-Mutis MC, Vreden S, Douine M. Implementation of a novel malaria management strategy based on self-testing and self-treatment in remote areas in the Amazon (Malakit): confronting a-priori assumptions with reality. BMC Public Health. 2022 Apr 15;22(1):770. doi: 10.1186/s12889-022-12801-0. PMID 35428230